CLINICAL TRIAL: NCT02076607
Title: Thoracic And Lumbar Burst Fracture: Correlation Between Structural Changes And Clinical Outcome Of Treatment
Status: Completed | Type: Observational
Sponsor: Hospital Ortopedico de Passo Fundo (Other)
Responsible Party: Principal Investigator, Diego da Silva Collares, Spinal surgery fellow, Hospital Ortopedico de Passo Fundo
Other Study IDs: 314151; 314151 (Registry Identifier: Fratura Explosão)
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Traumatic Burst Fractures of the Thoracic or Lumbar Spine.; Normal Neurological Function
Keywords: vertebra; column; lumbar; toracica; fracture; burst
MeSH Terms: conditions — Fractures, Bone | interventions — Arthrodesis; Braces

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conservative Treatment: Eleven patients underwent conservative treatment with Brace.
  Interventions: Device: Brace
- Surgical Treatment: Fourteen patients who underwent surgical treatment (arthrodesis).
  Interventions: Procedure: Arthrodesis

INTERVENTIONS:
Procedure: Arthrodesis — Posterior approach to toracolumbar spine fusion.
  Other Names: PLIF; TLIF
  Groups: Surgical Treatment
Device: Brace — Toracolumbar imobilization
  Other Names: Jewett; Putti
  Groups: Conservative Treatment

SUMMARY:
Evaluate the correlation between the structural changes of fractures of the thoracic and lumbar spine burst type with clinical outcome of the treatment.

DETAILED DESCRIPTION:
The treatment of burst fractures of the thoracic and lumbar spine is still a subject of much discussion and debate in the literature, especially in patients without neurological deficit. Most authors recommend surgical treatment for patients whose fracture shows signs of instability: 50% loss of vertebral body height, kyphosis with more than 30 degrees, involvement of more than 50% of the spinal canal. The authors advocate that this type of treatment uses the shorter hospital stay, early patient mobility, better kyphosis correction, the possibility of spinal canal decompression and prevention of neurological deterioration, as arguments in its favor.However, observational studies in patients without neurological deficit, showed no difference in long-term functional outcomes in patients with this type of injury, regardless of the type of treatment used (surgical or conservative). This study will express the clinical results and morphological changes of the thoracic and lumbar spine, at a minimum follow-up of 24 months, comparing the findings of the patients undergoing surgical treatment with those found in undergoing conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thoracic or lumbar burst fracture, without neurological lesion treated by the principal investigator of the study and periodically monitored in the Service of the researcher, Orthopedic Hospital of Passo Fundo, with minimum follow-up of 24 months fracture.

Exclusion Criteria:

* Patients with neurological deficit or who have left before 24 months the follow-up.

Ages: 22 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical treatment Group: 14 samples Conservative Treatment Group: 11 samples
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Clinical and radiological outcome after two years of follow up: Pain (VAS), deformity (degrees) and quality of life (SF36 questionary) | Over Two Years
  Retrospective review of medical records and imaging studies (radiographs and CT scans) of 30 patients without neurological deficit, with fractures of the thoracic and lumbar burst-type, in the archives of the Orthopedic Hospital of Passo Fundo, in the period between 2002 to 2011 submitted the clinical follow-up or post-operative periodical by the principal investigator of the study. The fractures, of the selected patients will be classified according to Magerl et al. (AO). Minimum follow-up is 24 months. It should be emphasized that all patients underwent at follow-up, the measurement of visual analog pain scale (VAS), the SF36 quality of life questionnaire, radiographic measurements of kyphosis, collapse and narrowing of the spinal canal. The clinical results obtained with conservative and surgical treatment will be compared and correlated with the morphological changes presented by the fractured vertebra.

CONTACTS AND LOCATIONS:
Overall Officials: Diego S Collares, MD, Principal Investigator — Hospital Ortopedico de Passo Fundo; Rodrigo A Tisot, MD, Study Director — Hospital Ortopedico de Passo Fundo; Andrius Berardi, MD, Principal Investigator — Hospital Ortopedico de Passo Fundo
Locations (1):
- Hospital Ortopedico de Passo Fundo, Passo Fundo, Rio Grande do Sul, Brazil